CLINICAL TRIAL: NCT04026438
Title: Randomized Controlled Trial to Study the Outcome of Intravenous Phosphate Supplementation in Live Donors Undergoing Hepatectomy for Living Donor Liver Transplantation (LDLT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Vivek Rajendran, Senior Resident, Department of HPB surgery and liver transplantation, Institute of Liver and Biliary Sciences, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ILBS-livertransplant
Record Dates: First submitted 2019-07-11; First posted 2019-07-19 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Complication, Postoperative; Regeneration Liver
MeSH Terms: conditions — Postoperative Complications | interventions — potassium phosphate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm - potassium phosphate injection (Experimental)
  Interventions: Drug: Potassium Phosphate Injection
- Control Arm (No Intervention)

INTERVENTIONS:
Drug: Potassium Phosphate Injection — One ml of the preparation contains 3 mmol of phosphorous which when equated with RDA 10ml ie 30 mmol of preparation will be supplemented. The preparation is given slowly, intravenously over 4 hours diluted in 500 ml normal saline
  Arms: Intervention Arm - potassium phosphate injection

SUMMARY:
In this study, we aim to analyse the effect of phosphate supplementation on donors undergoing partial hepatectomy for LDLT. In Group A, we are going to supplement phosphate in donors postoperatively from day 1 to day 5. We will analyse the trend of serum phosphate levels in donors postoperatively, its correlation with occurrence of postoperative complications and status of liver regeneration by CT volumetry on Day 7. Group B will constitute the controls for the study and hence attempt to find out the effect of phosphate supplementation in all donors postoperatively. We will analyse the data and elucidate the value of phosphate supplementation in reducing the occurrence of complications and effect on liver regeneration in donors in LDLT.

ELIGIBILITY:
Inclusion Criteria:

* All donors evaluated as per institutional protocol for donor hepatectomy and found fit
* Those who consent.

Exclusion Criteria:

* Patients refusing to consent for inclusion in the study.
* Minor hepatectomy
* Those who develop profound hypophosphatemia in the control group

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Post operative complications | 1 month
  Outcome of phosphate supplementation in reducing the occurrence of postoperative complications assessed by Clavien Dindo grading

SECONDARY OUTCOMES:
Trend of serum phosphorous levels | 1 week
  Serum phosphorous levels will be done daily and its trend will be compared in both the groups
Trends in post-operative liver function tests | 1 week
  Liver function tests will be done in both groups and its correlation with serum phosphate levels will be correlated
Duration of hospital, ICU stay | Till patient is discharged on an average of 10 days
  ICU stay and total hospital stay in the group will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Viniyendra Pamecha, Professor, Study Chair — Professor and Head, Department of HPB surgery and Liver transplantation, ILBS, New Delhi.
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided